CLINICAL TRIAL: NCT01869114
Title: A Phase II Study of Azacitidine and Sirolimus for the Treatment of High Risk Myelodysplastic Syndrome or Acute Myeloid Leukemia Refractory to or Not Eligible for Intensive Chemotherapy
Brief Title: Sirolimus and Azacitidine in Treating Patients With High Risk Myelodysplastic Syndrome or Acute Myeloid Leukemia That is Recurrent or Not Eligible for Intensive Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12D.587; 2012-50 (Other: CCRRC); JT 3016 (Other: JeffTrial Number)
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); de Novo Myelodysplastic Syndromes; Myelodysplastic Syndrome With Isolated Del(5q); Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Chromosome 5q Deletion Syndrome; Leukemia, Myeloid, Acute | interventions — Sirolimus; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High risk Myleodysplastic Syndrome (MDS) (Experimental): Patients receive sirolimus PO on days 1-10 or 1-12 and azacitidine IV on days 4-8, 11, and 12 or days 4-10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sirolimus; Drug: Azacitidine
- Acute Myeloid Leukemia (AML) (Experimental): Patients receive sirolimus PO on days 1-10 or 1-12 and azacitidine IV on days 4-8, 11, and 12 or days 4-10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sirolimus; Drug: Azacitidine
- MDS or AML with prior Azacitadine therapy (Experimental): Patients receive sirolimus PO on days 1-10 or 1-12 and azacitidine IV on days 4-8, 11, and 12 or days 4-10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sirolimus; Drug: Azacitidine

INTERVENTIONS:
Drug: Sirolimus — Given PO
  Other Names: rapamycin; Rapamune
Drug: Azacitidine — Given IV
  Other Names: 5-azacytidine; Vidaza

SUMMARY:
This phase II trial studies how well sirolimus and azacitidine works in treating patients with high-risk myelodysplastic syndrome or recurrent acute myeloid leukemia. Sirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Sirolimus and azacitidine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize the rate of response to azacitidine and sirolimus in adults with high-risk myelodysplastic syndrome (MDS), or relapsed or refractory acute myeloid leukemia (AML) or those unable or unwilling to tolerate high dose chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the pharmacodynamic effect of sirolimus on inhibition of mammalian target of rapamycin (mTOR) signaling in adults with high-risk MDS, or relapsed or refractory AML or those unable or unwilling to tolerate high dose chemotherapy.

II. To determine the safety and tolerability of sirolimus and azacitidine in adults with high-risk MDS, or relapsed or refractory AML or those unable or unwilling to tolerate high dose chemotherapy.

III. To determine the progression free survival and overall survival in adults with high-risk MDS, or relapsed or refractory AML or those unable or unwilling to tolerate high dose chemotherapy.

IV. To determine if the quality of life of patients is improved with the combination of azacitidine and sirolimus when compared to historical controls of azacitidine alone.

OUTLINE:

Patients receive sirolimus orally (PO) on days 1-10 or 1-12 and azacitidine intravenously (IV) on days 4-8, 11, and 12 or days 4-10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of one of the following:

   * MDS (Arm A): High-risk MDS defined as: >5% blasts in bone marrow and/or the following cytogenetic categories: presence of inv(3)/t(3q)/del(3q), -7/del(7q), complex cytogenetics (3 or more abnormalities)
   * AML (Arm B): Relapsed/refractory/unable to tolerate conventional chemotherapy
   * MDS or AML as above BUT with prior therapy with Azacitibine (Arm C): Patients who meet criteria for either Arm A or Arm B but have been treated or are currently treated with Azacitibine *Note: As of July 2018, only high risk MDS patients will be eligible as Arm B is closed. As of October 2017, those patients with MDS who have received prior treatment will now be enrolled in Arm A as Arm C is closed.
2. Patients must be ≥ 18 years old
3. Patients must have an ECOG performance status of <= 2 (see Attachment 1).
4. Patients must have a life expectancy of at least 4 weeks.
5. Patients must be able to consume oral medication.
6. Patients must have completed any radiotherapy four weeks prior to study entry, 0-2 weeks for local palliative XRT (small port).
7. Patients must have recovered from the toxic effects of any prior chemotherapy to < Grade 2 (except for alopecia).
8. Required initial laboratory values: Creatinine≤ 2.0mg/dL; total or direct bilirubin ≤ 1.5mg/dL (if not due to the leukemia itself or known Gilbert's Syndrome);(as documented by treating physician) SGPT(ALT) ≤ 3xULN; glucose <200 mg/dL, negative pregnancy test for women of child-bearing potential.
9. Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.
10. Patients may have had a prior stem cell transplant (autologous or allogeneic), however they may not have active GvHD, nor be on any immunosuppression

Exclusion Criteria:

1. Patients must not be receiving any chemotherapy agents (except Hydroxyurea)

   * Intrathecal ARA-C and intrathecal methotrexate are permissible (as they are not systemic and only isolated to the central nervous system).
   * Patients can not have received more than 3 prior lines of therapy for their hematologic malignancy. Patient may have previously had azacitidine or decitabine will be eligible to enroll on Arm A (MDS)
2. Patients must not be receiving growth factors.
3. Patients with a current second malignancy requiring systemic therapy, other than non-melanoma skin cancers, are not eligible. If a patient has had a prior second malignancy that is not currently requiring active treatment, the patient will be considered eligible.
4. Patients with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, myocardial infarction within the past 6 months or serious uncontrolled cardiac arrhythmia are not eligible.
5. Patients may not take any of the following medications while on study, but will be considered eligible if medication is discontinued 72 hrs prior to first dose of Sirolimus:

   * Carbamazepine (e.g. Tegretol)
   * Rifabutin (e.g. Mycobutin)
   * Rifampin (e.g. Rifadin)
   * Rifapentine (e.g. Priftin)
   * St. John's Wort- may decrease effects of sirolimus by decreasing the amount of sirolimus in the body
   * Clarithromycin (e.g. Biaxin)
   * Cyclosporin e.g. (Neoral or Sandimmune)
   * Diltiazem (e.g. Cardizem)
   * Erythromycin (e.g. Akne-Mycin, Ery-Tab)
   * Itraconazole (e.g. Sporanox)
   * Fluconazole (e.g. Diflucan)
   * Ketoconazole (e.g. Nizoral)
   * Telithromycin (e.g. Ketek)
   * Verapamil (e.g. Calan SR, Isoptin, Verelan)
   * Voriconazole (e.g. VFEND) - May increase the effects of sirolimus by increasing the amount of this medicine in the body. Can take 72 hours after last dose of Sirolimus
   * Tacrolimus (e.g. Prograf) - May cause liver transplant rejection or serious side effects in patients on sirolimus.
6. Patients with known HIV positivity or AIDS-related illness are not eligible.
7. Patients with other severe concurrent disease which in the judgment of the investigator would make the patient inappropriate for entry into this study are ineligible.
8. Patients must not have received any investigational agents within 21days of study entry.
9. Patients must not be pregnant or breastfeeding. Pregnancy tests must be obtained for all females of child-bearing potential. Pregnant or lactating patients are ineligible for this study due to the unknown human fetal or teratogenic toxicities of rapamycin. Males or females of reproductive age may not participate unless they have agreed to use an effective contraceptive method.
10. Patients who have uncontrolled infection are not eligible. Patients must have any active infections under control. Fungal disease must be stable for at least 2 weeks before study entry. Patients with bacteremia must have documented negative blood cultures prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kasner, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University
Locations (5):
- United States (5):
  - Jefferson Health NJ Division (Kennedy Hospital), Sewell, New Jersey
  - Abington Hospital - Jefferson Health, Abington, Pennsylvania
  - Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Jefferson Health, Aria Hospital, Philadelphia, Pennsylvania
  - Jefferson Health, Methodist Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Harris NL, Jaffe ES, Diebold J, Flandrin G, Muller-Hermelink HK, Vardiman J, Lister TA, Bloomfield CD. The World Health Organization classification of neoplastic diseases of the hematopoietic and lymphoid tissues. Report of the Clinical Advisory Committee meeting, Airlie House, Virginia, November, 1997. Ann Oncol. 1999 Dec;10(12):1419-32. doi: 10.1023/a:1008375931236. PMID 10643532
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Garcia-Manero G, Fenaux P. Hypomethylating agents and other novel strategies in myelodysplastic syndromes. J Clin Oncol. 2011 Feb 10;29(5):516-23. doi: 10.1200/JCO.2010.31.0854. Epub 2011 Jan 10. PMID 21220589
- [Background] Rollison DE, Howlader N, Smith MT, Strom SS, Merritt WD, Ries LA, Edwards BK, List AF. Epidemiology of myelodysplastic syndromes and chronic myeloproliferative disorders in the United States, 2001-2004, using data from the NAACCR and SEER programs. Blood. 2008 Jul 1;112(1):45-52. doi: 10.1182/blood-2008-01-134858. Epub 2008 Apr 28. PMID 18443215
- [Background] Silverman LR, Demakos EP, Peterson BL, Kornblith AB, Holland JC, Odchimar-Reissig R, Stone RM, Nelson D, Powell BL, DeCastro CM, Ellerton J, Larson RA, Schiffer CA, Holland JF. Randomized controlled trial of azacitidine in patients with the myelodysplastic syndrome: a study of the cancer and leukemia group B. J Clin Oncol. 2002 May 15;20(10):2429-40. doi: 10.1200/JCO.2002.04.117. PMID 12011120
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Jabbour E, Garcia-Manero G, Batty N, Shan J, O'Brien S, Cortes J, Ravandi F, Issa JP, Kantarjian H. Outcome of patients with myelodysplastic syndrome after failure of decitabine therapy. Cancer. 2010 Aug 15;116(16):3830-4. doi: 10.1002/cncr.25247. PMID 20564137
- [Background] Fenaux P, Gattermann N, Seymour JF, Hellstrom-Lindberg E, Mufti GJ, Duehrsen U, Gore SD, Ramos F, Beyne-Rauzy O, List A, McKenzie D, Backstrom J, Beach CL. Prolonged survival with improved tolerability in higher-risk myelodysplastic syndromes: azacitidine compared with low dose ara-C. Br J Haematol. 2010 Apr;149(2):244-9. doi: 10.1111/j.1365-2141.2010.08082.x. Epub 2010 Feb 5. PMID 20136825
- [Background] Cashen AF, Schiller GJ, O'Donnell MR, DiPersio JF. Multicenter, phase II study of decitabine for the first-line treatment of older patients with acute myeloid leukemia. J Clin Oncol. 2010 Feb 1;28(4):556-61. doi: 10.1200/JCO.2009.23.9178. Epub 2009 Dec 21. PMID 20026803
- [Background] Sudan N, Rossetti JM, Shadduck RK, Latsko J, Lech JA, Kaplan RB, Kennedy M, Gryn JF, Faroun Y, Lister J. Treatment of acute myelogenous leukemia with outpatient azacitidine. Cancer. 2006 Oct 15;107(8):1839-43. doi: 10.1002/cncr.22204. PMID 16967444
- [Background] Maurillo L, Venditti A, Spagnoli A, Gaidano G, Ferrero D, Oliva E, Lunghi M, D'Arco AM, Levis A, Pastore D, Di Renzo N, Santagostino A, Pavone V, Buccisano F, Musto P. Azacitidine for the treatment of patients with acute myeloid leukemia: report of 82 patients enrolled in an Italian Compassionate Program. Cancer. 2012 Feb 15;118(4):1014-22. doi: 10.1002/cncr.26354. Epub 2011 Jul 14. PMID 21761399
- [Background] Sun D, Toan X, Zhang Y, Chen Y, Lu R, Wang X, Fang J. Mammalian target of rapamycin pathway inhibition enhances the effects of 5-aza-dC on suppressing cell proliferation in human gastric cancer cell lines. Sci China C Life Sci. 2008 Jul;51(7):640-7. doi: 10.1007/s11427-008-0080-2. Epub 2008 Jul 13. PMID 18622747
- [Background] Zhang YJ, Zhao SL, Tian XQ, Sun DF, Xiong H, Dai Q, Li XQ, Fang JY. Combined inhibition of Dnmt and mTOR signaling inhibits formation and growth of colorectal cancer. Int J Colorectal Dis. 2009 Jun;24(6):629-39. doi: 10.1007/s00384-009-0664-8. Epub 2009 Feb 20. PMID 19229543
- [Background] Wei AH, Tan PT, Catalano J, et al. Azacitidine in Combination with the mTOR Inhibitor Everolimus in Relapsed and Refractory AML. ASH Annual Meeting Abstracts. 2011;118:2599.
- [Background] Morris RE. Rapamycin: FK506's fraternal twin or distant cousin? Immunol Today. 1991 May;12(5):137-40. doi: 10.1016/S0167-5699(05)80040-4. PMID 1715165
- [Background] Brown VI, Fang J, Alcorn K, Barr R, Kim JM, Wasserman R, Grupp SA. Rapamycin is active against B-precursor leukemia in vitro and in vivo, an effect that is modulated by IL-7-mediated signaling. Proc Natl Acad Sci U S A. 2003 Dec 9;100(25):15113-8. doi: 10.1073/pnas.2436348100. Epub 2003 Dec 1. PMID 14657335
- [Background] Gottschalk AR, Boise LH, Thompson CB, Quintans J. Identification of immunosuppressant-induced apoptosis in a murine B-cell line and its prevention by bcl-x but not bcl-2. Proc Natl Acad Sci U S A. 1994 Jul 19;91(15):7350-4. doi: 10.1073/pnas.91.15.7350. PMID 7518929
- [Background] Hultsch T, Martin R, Hohman RJ. The effect of the immunophilin ligands rapamycin and FK506 on proliferation of mast cells and other hematopoietic cell lines. Mol Biol Cell. 1992 Sep;3(9):981-7. doi: 10.1091/mbc.3.9.981. PMID 1384815
- [Background] Majewski M, Korecka M, Kossev P, Li S, Goldman J, Moore J, Silberstein LE, Nowell PC, Schuler W, Shaw LM, Wasik MA. The immunosuppressive macrolide RAD inhibits growth of human Epstein-Barr virus-transformed B lymphocytes in vitro and in vivo: A potential approach to prevention and treatment of posttransplant lymphoproliferative disorders. Proc Natl Acad Sci U S A. 2000 Apr 11;97(8):4285-90. doi: 10.1073/pnas.080068597. PMID 10759564
- [Background] Muthukkumar S, Ramesh TM, Bondada S. Rapamycin, a potent immunosuppressive drug, causes programmed cell death in B lymphoma cells. Transplantation. 1995 Aug 15;60(3):264-70. doi: 10.1097/00007890-199508000-00010. PMID 7544036
- [Background] Xu Q, Simpson SE, Scialla TJ, Bagg A, Carroll M. Survival of acute myeloid leukemia cells requires PI3 kinase activation. Blood. 2003 Aug 1;102(3):972-80. doi: 10.1182/blood-2002-11-3429. Epub 2003 Apr 17. PMID 12702506
- [Background] Yamamoto-Yamaguchi Y, Okabe-Kado J, Kasukabe T, Honma Y. Induction of differentiation of human myeloid leukemia cells by immunosuppressant macrolides (rapamycin and FK506) and calcium/calmodulin-dependent kinase inhibitors. Exp Hematol. 2001 May;29(5):582-8. doi: 10.1016/s0301-472x(01)00626-9. PMID 11376870
- [Background] Xu Q, Thompson JE, Carroll M. mTOR regulates cell survival after etoposide treatment in primary AML cells. Blood. 2005 Dec 15;106(13):4261-8. doi: 10.1182/blood-2004-11-4468. Epub 2005 Sep 8. PMID 16150937
- [Background] Perl AE, Kasner MT, Tsai DE, Vogl DT, Loren AW, Schuster SJ, Porter DL, Stadtmauer EA, Goldstein SC, Frey NV, Nasta SD, Hexner EO, Dierov JK, Swider CR, Bagg A, Gewirtz AM, Carroll M, Luger SM. A phase I study of the mammalian target of rapamycin inhibitor sirolimus and MEC chemotherapy in relapsed and refractory acute myelogenous leukemia. Clin Cancer Res. 2009 Nov 1;15(21):6732-9. doi: 10.1158/1078-0432.CCR-09-0842. Epub 2009 Oct 20. PMID 19843663
- [Background] Zeng Z, Sarbassov dos D, Samudio IJ, Yee KW, Munsell MF, Ellen Jackson C, Giles FJ, Sabatini DM, Andreeff M, Konopleva M. Rapamycin derivatives reduce mTORC2 signaling and inhibit AKT activation in AML. Blood. 2007 Apr 15;109(8):3509-12. doi: 10.1182/blood-2006-06-030833. Epub 2006 Dec 19. PMID 17179228
- [Background] Atkins MB, Hidalgo M, Stadler WM, Logan TF, Dutcher JP, Hudes GR, Park Y, Liou SH, Marshall B, Boni JP, Dukart G, Sherman ML. Randomized phase II study of multiple dose levels of CCI-779, a novel mammalian target of rapamycin kinase inhibitor, in patients with advanced refractory renal cell carcinoma. J Clin Oncol. 2004 Mar 1;22(5):909-18. doi: 10.1200/JCO.2004.08.185. PMID 14990647
- [Background] Yee KW, Zeng Z, Konopleva M, Verstovsek S, Ravandi F, Ferrajoli A, Thomas D, Wierda W, Apostolidou E, Albitar M, O'Brien S, Andreeff M, Giles FJ. Phase I/II study of the mammalian target of rapamycin inhibitor everolimus (RAD001) in patients with relapsed or refractory hematologic malignancies. Clin Cancer Res. 2006 Sep 1;12(17):5165-73. doi: 10.1158/1078-0432.CCR-06-0764. PMID 16951235
- [Background] Teachey DT, Obzut DA, Cooperman J, Fang J, Carroll M, Choi JK, Houghton PJ, Brown VI, Grupp SA. The mTOR inhibitor CCI-779 induces apoptosis and inhibits growth in preclinical models of primary adult human ALL. Blood. 2006 Feb 1;107(3):1149-55. doi: 10.1182/blood-2005-05-1935. Epub 2005 Sep 29. PMID 16195324
- [Background] Vignot S, Faivre S, Aguirre D, Raymond E. mTOR-targeted therapy of cancer with rapamycin derivatives. Ann Oncol. 2005 Apr;16(4):525-37. doi: 10.1093/annonc/mdi113. Epub 2005 Feb 22. PMID 15728109
- [Background] Punt CJ, Boni J, Bruntsch U, Peters M, Thielert C. Phase I and pharmacokinetic study of CCI-779, a novel cytostatic cell-cycle inhibitor, in combination with 5-fluorouracil and leucovorin in patients with advanced solid tumors. Ann Oncol. 2003 Jun;14(6):931-7. doi: 10.1093/annonc/mdg248. PMID 12796032
- [Background] Witzig TE, Geyer SM, Ghobrial I, Inwards DJ, Fonseca R, Kurtin P, Ansell SM, Luyun R, Flynn PJ, Morton RF, Dakhil SR, Gross H, Kaufmann SH. Phase II trial of single-agent temsirolimus (CCI-779) for relapsed mantle cell lymphoma. J Clin Oncol. 2005 Aug 10;23(23):5347-56. doi: 10.1200/JCO.2005.13.466. Epub 2005 Jun 27. PMID 15983389
- [Background] Jennings CD, Foon KA. Recent advances in flow cytometry: application to the diagnosis of hematologic malignancy. Blood. 1997 Oct 15;90(8):2863-92. No abstract available. PMID 9376567
- [Background] Irish JM, Hovland R, Krutzik PO, Perez OD, Bruserud O, Gjertsen BT, Nolan GP. Single cell profiling of potentiated phospho-protein networks in cancer cells. Cell. 2004 Jul 23;118(2):217-28. doi: 10.1016/j.cell.2004.06.028. PMID 15260991
- [Background] Jacobberger JW, Sramkoski RM, Frisa PS, Ye PP, Gottlieb MA, Hedley DW, Shankey TV, Smith BL, Paniagua M, Goolsby CL. Immunoreactivity of Stat5 phosphorylated on tyrosine as a cell-based measure of Bcr/Abl kinase activity. Cytometry A. 2003 Aug;54(2):75-88. doi: 10.1002/cyto.a.10063. PMID 12879454
- [Background] Perez OD, Nolan GP. Simultaneous measurement of multiple active kinase states using polychromatic flow cytometry. Nat Biotechnol. 2002 Feb;20(2):155-62. doi: 10.1038/nbt0202-155. PMID 11821861
- [Background] Krutzik PO, Irish JM, Nolan GP, Perez OD. Analysis of protein phosphorylation and cellular signaling events by flow cytometry: techniques and clinical applications. Clin Immunol. 2004 Mar;110(3):206-21. doi: 10.1016/j.clim.2003.11.009. PMID 15047199
- [Background] Chow S, Hedley D, Grom P, Magari R, Jacobberger JW, Shankey TV. Whole blood fixation and permeabilization protocol with red blood cell lysis for flow cytometry of intracellular phosphorylated epitopes in leukocyte subpopulations. Cytometry A. 2005 Sep;67(1):4-17. doi: 10.1002/cyto.a.20167. PMID 16080188
- [Background] Chow S, Minden MD, Hedley DW. Constitutive phosphorylation of the S6 ribosomal protein via mTOR and ERK signaling in the peripheral blasts of acute leukemia patients. Exp Hematol. 2006 Sep;34(9):1183-91. doi: 10.1016/j.exphem.2006.05.002. PMID 16939811
- [Background] Hedley DW, Chow S, Goolsby C, Shankey TV. Pharmacodynamic monitoring of molecular-targeted agents in the peripheral blood of leukemia patients using flow cytometry. Toxicol Pathol. 2008 Jan;36(1):133-9. doi: 10.1177/0192623307310952. PMID 18337231
- [Background] Tong FK, Chow S, Hedley D. Pharmacodynamic monitoring of BAY 43-9006 (Sorafenib) in phase I clinical trials involving solid tumor and AML/MDS patients, using flow cytometry to monitor activation of the ERK pathway in peripheral blood cells. Cytometry B Clin Cytom. 2006 May;70(3):107-14. doi: 10.1002/cyto.b.20092. PMID 16498671
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Acute Myeloid Leukemia (AML); Arm B: High risk Myleodysplastic Syndrome (MDS): Patients receive sirolimus PO on days 1-10 or 1-12 and azacitidine IV on days 4-8, 11, and 12 or days 4-10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Sirolimus: Given PO
  Azacitidine: Given IV
- Arm C: MDS or AML with prior Azacitadine therapy: Patients receive sirolimus PO on days 1-10 or 1-12 and azacitidine IV on days 4-8, 11, and 12 or days 4-10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A: Acute Myeloid Leukemia (AML) | Arm B: High risk Myleodysplastic Syndrome (MDS) | Arm C: MDS or AML with prior Azacitadine therapy
Started | 21 | 28 | 8
Completed | 2 | 4 | 0
Not Completed | 19 | 24 | 8
Not completed — Death | 19 | 18 | 8
Not completed — Adverse Event/Side Effects/Complications | 0 | 1 | 0
Not completed — Patient off treatment for other complicating disease | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Disease Progression | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Acute Myeloid Leukemia (AML) | Arm B: High Risk Myleodysplastic Syndrome (MDS) | Arm C: MDS or AML With Prior Azacitadine Therapy | Total
Number analyzed (Participants) | 21 | 28 | 8 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 0 | 11
  >=65 years | 14 | 24 | 8 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 1 | 18
  Male | 13 | 19 | 7 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 19 | 24 | 8 | 51
  Unknown or Not Reported | 2 | 2 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 5 | 2 | 7
  White | 18 | 19 | 6 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 21 | 28 | 8 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: MDS: Patients meeting an erythroid response, a platelet response, or a neutrophil response will be considered responders.
  AML: Patients achieving a complete remission (CR), complete response in the absence of a total platelet recovery (CRp), or partial remission (PR) will be considered responders.
Time Frame: Up to 5 years
Population: Arm C was included in the study design, and eight participants were enrolled. However, none of them received study treatment, and no safety or efficacy data were collected. As a result, there is no evaluable data available for this outcome measure, and no data will be available in the future.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Acute Myeloid Leukemia (AML) | Arm B: High risk Myleodysplastic Syndrome (MDS) | Arm C: MDS or AML with prior Azacitadine therapy
Number analyzed (Participants) | 21 | 28 | 0
Participants
  Complete Response (CR) | 1 | 4 |
  Partial Response (PR) | 5 | 3 |
  Stable Disease (SD) | 13 | 6 |
  Progressive Disease (PD) | 4 | 4 |

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be assessed and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0. All AEs will be recorded and summarized by frequency and severity.
Time Frame: From the first dose of study drug through 30 days after the last dose of study treatment, an average of 7 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Acute Myeloid Leukemia (AML) | Arm B: High risk Myleodysplastic Syndrome (MDS) | Arm C: MDS or AML with prior Azacitadine therapy
Number analyzed (Participants) | 21 | 28 | 0
Participants | 20 | 11 |

3. Secondary Outcome: Mean Percentage of pS6-positive Blasts as Measured by Intracellular Flow Cytometry
Description: The mean percentage of pS6-positive blasts in bone marrow samples was measured using intracellular flow cytometry before and after sirolimus administration. A reduction in pS6-positive blasts indicates inhibition of mTOR signaling. Results are reported as mean values along with the corresponding range.
Time Frame: Up to day 4 before azacitidine administration
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Arm A: Acute Myeloid Leukemia (AML) | Arm B: High risk Myleodysplastic Syndrome (MDS) | Arm C: MDS or AML with prior Azacitadine therapy
Number analyzed (Participants) | 15 | 12 | 0
percentage change | 18.6 [4.4 to 49] | 37 [8 to 96] |

4. Secondary Outcome: Quality of Life (QOL) Assessed by the European Organization for Research and Treatment of Cancer (EORTC) QOL and the Mental Health Inventory (MHI)
Description: EORTC QOL a 30-item questionnaire covering functional scales, symptom scales, and a global health status/QOL scale. MHI is a validated patient-reported outcome instrument used to assess psychological well-being across multiple domains. Participants rate items on a 6-point Likert scale. Scores are transformed to a 0-100 scale, with higher scores indicated better mental health.
Time Frame: Up to day 164
Population: QoL questionnaire score analysis was contingent on demonstrating efficacy in the primary endpoint. The study did not met the primary efficacy endpoint, and QoL assessment was not performed as further data collection for secondary endpoints was not pursued.
Arm/Group | Arm A: Acute Myeloid Leukemia (AML) | Arm B: High risk Myleodysplastic Syndrome (MDS) | Arm C: MDS or AML with prior Azacitadine therapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The study period during which adverse events must be reported is normally defined as the period from the initiation of any study procedures to the end of the study treatment follow-up. For this study, the study treatment follow-up is defined as from the first dose of study drug through 30 days after the last dose of study treatment, an average of 7 months.
Description: All participant deaths are included in the All-Cause Mortality table. Deaths outside the prespecified AE collection window are excluded from the AE/SAE summary but fully represented in the mortality table.
Arm/Group | Arm A: Acute Myeloid Leukemia (AML) | Arm B: High risk Myleodysplastic Syndrome (MDS) | Arm C: MDS or AML With Prior Azacitadine Therapy
All-Cause Mortality (participants affected / at risk) | 19/21 | 18/28 | 0/8
Serious Adverse Events (participants affected / at risk) | 8/21 | 1/28 | 0/8
Other Adverse Events (participants affected / at risk) | 20/21 | 11/28 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Acute Myeloid Leukemia (AML) (N=21) | Arm B: High risk Myleodysplastic Syndrome (MDS) (N=28) | Arm C: MDS or AML With Prior Azacitadine Therapy (N=8)
Multi-organ failure (General disorders) | 2 (2) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) — Progressive Disease
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Acute Myeloid Leukemia (AML) (N=21) | Arm B: High risk Myleodysplastic Syndrome (MDS) (N=28) | Arm C: MDS or AML With Prior Azacitadine Therapy (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (4) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Vitreous Tear
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (15) | 5 (5) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 5 (7) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 5 (9) | 2 (4) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Infusion Related Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 7 (7) | 3 (3) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
skin infection- cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT01869114/Prot_SAP_000.pdf